CLINICAL TRIAL: NCT07336888
Title: A Study on the Application of Positive Psychological Counseling Based on "Dou Bao" Software in Patients With Post-stroke Depression
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Fourth Affiliated Hospital of Zhejiang University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KY-2025-303
Record Dates: First submitted 2025-12-04; First posted 2026-01-13 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2025-12

CONDITIONS: Stroke; Post Stroke Depression
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Doubao Software Group Application Team (Experimental): Utilize an active psychological counseling platform based on the "Doubao" software
  Interventions: Other: The positive psychological counseling platform of the "Doubao" software
- Conventional control group (No Intervention): Standard psychological care plan

INTERVENTIONS:
Other: The positive psychological counseling platform of the "Doubao" software — Utilize an active psychological counseling platform based on the "Doubao" software
  Arms: Doubao Software Group Application Team

SUMMARY:
Patients with PSD have the characteristics of high incidence rate, difficult identification and great harm. However, the existing AI chat platforms have not developed any relevant software or programs for PSD patients. Given that the chatbot function in the "Douba" software is relatively mature and can flexibly modify the corresponding intelligent agent according to user needs, this study intends to appropriately supplement and optimize the AI agent in the "Douba" software to explore the effect of the chatbot in the software in alleviating the symptoms of PSD patients.

ELIGIBILITY:
Inclusion Criteria:

* Meets the criteria of either the "Chinese Guidelines for the Diagnosis and Treatment of Acute Ischemic Stroke" or the "Chinese Guidelines for the Diagnosis and Treatment of Acute Cerebral Hemorrhage" and is confirmed by CT or MRI;
* Patients with stable vital signs and conditions;
* Meets the "Third Edition of the Classification and Diagnosis Criteria for Mental Disorders in China" and has a score of ≥5 on the 9-item Patient Health Questionnaire (PHQ-9) scale;
* Patients are over 18 years old;
* Can understand the relevant content of the scale correctly and provide answers independently or with the help of others, have clear consciousness and sign the consent form;
* Can use smartphones.

Exclusion Criteria:

* Those with severe functional impairments of important organs such as the heart, lungs, liver and kidneys;
* Those without a smart phone;

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2027-01-01 (Estimated); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Depression assessment | Before the intervention and 3 months after the intervention
  Use the PHQ-9 scale,The sensitivity of this scale in diagnosing depression was 0.82, and the specificity was 0.87. The PHQ-9 scale collects information on the degree to which the evaluated individuals are troubled by different depressive symptoms, including loss of interest, low mood, sleep disorders, feeling tired, changes in appetite, poor self-perception, lack of concentration, slow movements or irritability, and suicidal thoughts. The score for each item ranges from 0 (none at all) to 3 (almost every day), and the total score ranges from 0 to 27. The higher the score, the more severe the symptoms.

SECONDARY OUTCOMES:
appraisal of life quality | Before the intervention and 3 months after the intervention
  The assessment was conducted using the short version of the stroke-specific quality of life scale (SV-SS-QoL). This scale consists of 2 dimensions and 12 items. Each item is scored using the Likert 5-point scale, with values ranging from 1 to 5. The total score ranges from 12 to 60. A higher scale score indicates better quality of life. The Cronbach's α coefficient of this scale is 0.882, the split-half reliability is 0.845, and the test-retest reliability is 0.839.
the satisfaction of patients | 3 months after the intervention
  Have the patients rate their satisfaction with the psychological counseling method used in this study on a scale of 1 to 5. If they feel extremely dissatisfied, they should give a score of 1; if they are dissatisfied, 2; if they are basically satisfied, 3; if they are moderately satisfied, 4; and if they feel extremely satisfied, 5. For those who give a score of extremely dissatisfied or extremely satisfied, ask them for the specific reasons to prevent them from giving random scores.
Research dropout rate | 3 months after the intervention
  After comparing the two groups of patients 3 months later, the study withdrawal rates were determined. The study withdrawal rate = the number of people in this group 3 months later / the initial number of people in this group in the study × 100%.

IPD SHARING:
Plan to Share IPD: No